CLINICAL TRIAL: NCT04261569
Title: Clinical Trial for Near Infrared Endoventricular Illumination for Neuroprotection in Very Early Cases of Parkinson's Disease (Ev-NIRT)
Acronym: Ev-NIRT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Collaborators: Commissariat A L'energie Atomique (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 38RC19.098; 2019-A02097-50 (Other: ANSM ID RCB)
Record Dates: First submitted 2020-01-27; First posted 2020-02-10 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Very Early Stage of Parkinson's Disease
Keywords: Parkinson's disease (PD); Intraventricular illumination by near-infrared light (Ev-NIRT); Positron Emission Tomography (PET); Substantia Nigra Pars Compacta (SNpc); Photobiomodulation; Medical Device (MD)
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Intervention Model Description: One control arm : patients without any medical device One illuminated arm : patients with intraventricular near-infrared light illumination
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Illuminated arm (Experimental): patients with intraventricular near-infrared light illumination
  Interventions: Device: Ev-NIRT
- control arm (No Intervention): patients without any medical device

INTERVENTIONS:
Device: Ev-NIRT — Endoventricular near infra red treatment : Intraventricular pulsed, chronic, cyclic, near-infrared illumination of the Central Nervous System (CNS) at 150 Hz, 15 mW, 1 minute ON and 5 minutes OFF
  Arms: Illuminated arm

SUMMARY:
Parkinson's disease has only pharmacological (essentially dopaminergic) and surgical treatment (essentially high-frequency deep brain stimulation), that are symptomatically effective. none of them is curative, and has the ability to slow down the disease and to protect dopaminergic neurons from death by neurodegeneration. Experimental results, based on preclinical studies, suggest that brain illumination in the Near-InfraRed (NIR) range is likely to slow down this neurodegenerative process.

Thus, a medical device system (called Ev-NIRT) has been developed for 670 nm intracerebral illumination of the substantia nigra pars compacta (SNpc), and is planned to be tested for the treatment of Parkinson's disease.

In this pilot study the investigators will evaluate the feasibility and tolerance of surgery and brain illumination thanks to the Ev-NIRT medical device, in a group of 7 de novo Parkinson's patients implanted with the innovative medical device. Patients will be monitored for 4 years.

DETAILED DESCRIPTION:
The level of neuroprotection induced by illumination at 670nm appears effective in preclinical studies, and justify the transfer into a clinical trial. The investigators currently have developed and produced implantable devices, to be implanted into the brain through a minimally invasive endoventricular route. The electrical energy required is supplied by the batteries adapted from those used for deep brain stimulation.

The feasibility of trans ventricular implantation is ensured by the experience gained by our team in the endoventricular stimulation of the posterior hypothalamus in the cluster headache.

In this clinical study, the investigators will evaluate the tolerance and safety of intraventricular surgical technic and illumination by the Ev-NIRT medical device implanted into the brain of 7 patients with Parkinson's disease. idiopathic, aged 25-65 years, at a very early stage (less than 2 years of evolution). The NIR illumination will begin immediately after surgery.

The investigators will also evaluate secondarily, the neuroprotective effect of this new treatment modality, by comparing the decrease of dopaminergic neurons by Positron Emission Tomography (PET)-scan using [11C]PE2I) tracer of implanted patients to that of a control group of 7 patients whose characteristics in terms of duration of evolution and clinical severity are identical, but who are not implanted, and therefore not exposed to NIR illumination.

The PET-scan-PE2I exam is conducted in both groups annually for 4 years (a total of 5 measurements) and compared to the PE2I PET obtained at the beginning of participation in the study. A group-wide comparison will be made between the NIR group and the control group.

ELIGIBILITY:
Inclusion Criteria:

1. Clinically diagnosed idiopathic Parkinson's disease according to MDS criteria developed by R.B. Postuma (Anang et al, Neurology, 2014)
2. Dopaminergic denervation confirmed in PET [11C]PE2I with a decrease in tracer fixation at the striatum level of at least 30% on average compared to the white matter fixation of the cerebellum
3. Patients willing to start dopaminergic treatment
4. Very early stage of the disease:

   1. Diagnosis of recent Parkinson's disease (less than two years after a neurologist's diagnosis)
   2. Hoehn and Yahr Stage 1 to 2
   3. Maximum 2 tremor on the MDS-UPDRS scale
   4. Naive of any anti-Parkinsonian treatment
5. Between 25 and 65 years of age
6. Score on Beck Depression Inventory (BDI) scale below the value of 20
7. Easy handling of the French language in oral and written language
8. Social security affiliates or beneficiaries of such a scheme
9. Informed and written consent signed by the patient

Exclusion Criteria:

1. All categories of protected persons: pregnant woman, parturient, breastfeeding mother, person deprived of liberty by judicial or administrative decision, person subject to a measure of legal protection, hospitalized for psychiatric disorder
2. Carcinological history in the previous 5 years, not stabilized
3. Uncontrolled medical condition that may lead to complications
4. Preoperative brain Magnetic Resonance Imaging (MRI) showing brain damage that may be responsible for Parkinson's syndrome or a significant surgical risk (e.g. vascular malformation)
5. Surgical or anesthetic contraindication
6. History of brain infection with herpes virus
7. Contraindication to MRI (claustrophobia, non-compatible mri metal prosthesis, etc.)
8. Predictable need for frequent use of MRI scans after surgery
9. Unstabilized psychotropic treatment
10. Patient with cognitive impairment at the outset of illness (Montreal Cognitive Assessment (MoCA) score - 26)
11. Atypias suspecting atypical Parkinson's syndrome
12. Chronic treatment with L-Dopa or dopamine agonist
13. Presence of another serious pathology (major depressive episode, suicidal patient, active psychosis ...)
14. Participation in another interventional clinical trial
15. Wearing pace makers other than brain

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Estimated)
Dates: Start 2020-12-14 (Actual); Primary Completion 2029-01 (Estimated); Study Completion 2032-04 (Estimated)

PRIMARY OUTCOMES:
Incidence of Ev-NIRT Treatment on Emergent Adverse Events (Tolerance) after surgical intervention and NIR illumination following the implantation of the Ev-NIRT medical device | 4 years
  Emergent Adverse Events [Safety and Tolerability]

SECONDARY OUTCOMES:
Characterization of annual neuronal loss observed by decrease in tracer fixation at the striatum level | 4 years
  Annual measurement of dopaminergic denervation in Positron Emission Tomography (PET) using [11C]PE2I tracer fixation at the striatum level in percentage compared to the white matter fixation of the cerebellum
Evaluation of the motor clinical signs progression | 4 years
  Scores on the Movement Disorder Society-Sponsored Revision of the Unified Parkinson's Disease Rating Scale (MDS-UPDRS scale sections II, III and IV) [0-100% : higher scores mean worse outcome]
Evaluation of the non-motor bahavioral signs progression | 4 years
  Scores on the non-motor scales Behavioral Evaluation in Parkinson's disease (ECMP) [0-4 : higher scores mean worse outcome]
Evaluation of the non-motor clinical signs progression | 4 years
  Scores on the non-motor scales Lille Apathy Rating Scale (LARS) [-4/+4 : higher scores mean worse outcome]
Evaluation of depression signs progression | 4 years
  Scores on the non-motor scales Beck Depression Inventory (BDI-II) [0-3 : higher scores mean worse outcome]
Evaluation of the non-motor symptoms signs progression | 4 years
  Scores on the non-motor scales Non Motor Symptoms scale (NMS) [0-30 : higher scores mean better outcome]
Comparison between the date of diagnosis and the date of introduction of substitution therapy with dopaminergic drugs or dopamine agonists | 4 years
  Time period between the date of diagnosis and the date of introduction of dopaminergic substitute therapy or dopaminergic agonists
Evolution of this prescription of substitution therapy over the duration of study | 4 years
  Follow up of dosage of dopaminergic substitute therapy or dopaminergic agonists
Assessment in both groups of the time it takes for the onset of different motor symptoms (including tremor, akinesia and stiffness, speech, walking and balance disorders) and not motor symptoms of Parkinson's disease in relation to initial diagnosis. | 4 years
  Time period between the date of diagnosis and the date of onset of different motor and non-motor symptoms objectified by an increase in item scores specific to these symptoms on the Movement Disorder Society-Sponsored Revision of the Unified Parkinson's Disease Rating Scale (MDS-UPDRS scale) passed into OFF drug [0-100% : higher scores mean worse outcome]
Evolution of the quality of life of patients in both groups | 4 years
  Parkinson Disease Quotation (PDQ-39) quiz score [0-4 : higher scores mean worse outcome]
Evolution of walking speed in both patient groups | 4 years
  Right and left foot speed measured during a walking task on the Vicon platform without and with dopaminergic treatment
Evolution of walking parameters in both patient groups | 4 years
  Score in the "freezing of gait" questionnaire [0-24 : higher scores mean worse outcome] without and with dopaminergic treatment

CONTACTS AND LOCATIONS:
Overall Officials: Stephan CHABARDES, MD, PhD, Principal Investigator — University Hospital, Grenoble
Locations (1):
- CLINATEC, Grenoble, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chabardes S, Carron R, Seigneuret E, Torres N, Goetz L, Krainik A, Piallat B, Pham P, David O, Giraud P, Benabid AL. Endoventricular Deep Brain Stimulation of the Third Ventricle: Proof of Concept and Application to Cluster Headache. Neurosurgery. 2016 Dec;79(6):806-815. doi: 10.1227/NEU.0000000000001260. PMID 27244468
- [Background] Darlot F, Moro C, El Massri N, Chabrol C, Johnstone DM, Reinhart F, Agay D, Torres N, Bekha D, Auboiroux V, Costecalde T, Peoples CL, Anastascio HD, Shaw VE, Stone J, Mitrofanis J, Benabid AL. Near-infrared light is neuroprotective in a monkey model of Parkinson disease. Ann Neurol. 2016 Jan;79(1):59-75. doi: 10.1002/ana.24542. Epub 2015 Dec 12. PMID 26456231
- [Background] Moro C, El Massri N, Darlot F, Torres N, Chabrol C, Agay D, Auboiroux V, Johnstone DM, Stone J, Mitrofanis J, Benabid AL. Effects of a higher dose of near-infrared light on clinical signs and neuroprotection in a monkey model of Parkinson's disease. Brain Res. 2016 Oct 1;1648(Pt A):19-26. doi: 10.1016/j.brainres.2016.07.005. Epub 2016 Jul 7. PMID 27396907
- [Background] Reinhart F, Massri NE, Chabrol C, Cretallaz C, Johnstone DM, Torres N, Darlot F, Costecalde T, Stone J, Mitrofanis J, Benabid AL, Moro C. Intracranial application of near-infrared light in a hemi-parkinsonian rat model: the impact on behavior and cell survival. J Neurosurg. 2016 Jun;124(6):1829-41. doi: 10.3171/2015.5.JNS15735. Epub 2015 Nov 27. PMID 26613166
- [Background] Johnstone DM, Moro C, Stone J, Benabid AL, Mitrofanis J. Turning On Lights to Stop Neurodegeneration: The Potential of Near Infrared Light Therapy in Alzheimer's and Parkinson's Disease. Front Neurosci. 2016 Jan 11;9:500. doi: 10.3389/fnins.2015.00500. eCollection 2015. PMID 26793049